CLINICAL TRIAL: NCT04090437
Title: Dipole Intracardiac Mapping With ACUTUS System for Catheter Ablation of Atrial Fibrillation in Hypertrophic Cardiomyopathy
Brief Title: HCM-AF Ablation With ACUTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUTUS-RBH01
Record Dates: First submitted 2019-09-05; First posted 2019-09-16 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Atrial Fibrillation; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Prospective, double-arm, randomised, observational study that will recruit 20 HCM-AF patients (10 for each group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 - PVI first step (Active Comparator): Catheter ablation procedure:
  Dipole map of RA and LA at baseline (5 times for both, each for 20sec, +/- Adenosine IV)
  * PVI as first step
  * Remap to assess any change in activation
  * Ablate all rotors (API) in LA until SR or DCCV
  * Deployment of RA CTI line and demonstration of bidirectional block
  Interventions: Procedure: Catheter ablation procedure
- Group2 - PVI last step (Active Comparator): Catheter ablation procedure:
  Dipole map of RA and LA at baseline (5 times for both, each for 20sec, +/- Adenosine IV)
  * Ablate all rotors (API) in LA until SR or DCCV
  * Remap to assess any change in activation
  * PVI as last step even when SR achieved earlier
  * Deployment of RA CTI line and demonstration of bidirectional block
  Interventions: Procedure: Catheter ablation procedure

INTERVENTIONS:
Procedure: Catheter ablation procedure — Catheter ablation procedure using Acutus mapping system

SUMMARY:
BACKGROUND About 1/4 of patients with hypertrophic cardiomyopathy (HCM) seem to develop atrial fibrillation (AF) over their life-span. Typically, symptoms of heart failure and especially shortness of breath get much worse once AF is present. Catheter ablation of AF in HCM has been proposed by several centres, but outcomes are much worse than in non-HCM AF. Accurate mapping of the arrhythmia is crucial with regard to improving the procedural outcome. Interestingly, intracardiac mapping during AF has demonstrated very long average cycle length during ongoing AF in HCM which should make identification of the critical re-entry/rotors much easier using dipole cardiac mapping (Acutus mapping system, Acutus Medical, CA, USA).

POPULATION and PURPOSE This is a pilot trial recruiting a total of 20 patients with HCM and AF (paroxysmal or persistent with <12 months duration time in persistent AF) eligible for catheter ablation, without other significant structural heart disease Primary endpoints

Safety:

* Absence of acute adverse events due to the use of ACUTUS mapping system during AF ablation
* Evidence of chronic adverse events due to the use of ACUTUS mapping system guided catheter ablation during the 12 months F/U period
* Safety endpoint of the entire mapping and ablation strategy

Efficacy:

* Assessment on efficacy of ACUTUS mapping system guided AF ablation in HCM patients using a double-arm study design
* RF time to termination of AF to SR Secondary endpoints
* RF time to termination of AF to atrial tachycardia (AT)
* Freedom from AF/flutter/tachycardia (> 30 sec) at the end of the 12 months follow up (F/U) period
* Time to first recurrence of AF/flutter/tachycardia (> 30 sec)
* Freedom of AF/flutter/tachycardia on previously failed anti-arrhythmic medication Ablation procedure First 10 patients (group 1): ablation will be carried out after acquisition of a left atrium (LA) and right atrium (RA) dipole map at baseline, pre and post administration of Adenosine IV. Then pulmonary vein isolation (PVI) as a first step and subsequent remap and ablation of all patterns of interest in the LA until restoration of sinus rhythm (SR) or decision to proceed with direct current cardioversion (DCCV, 360J).

Second 10 patients (group 2): after the acquisition of a dipole map of LA and RA at baseline (pre and post Adenosine IV administration), ablation of all identified areas of interest (API) will be performed, followed by remap and finally PVI +/- DCCV.

For all patients: final step will be the deployment of a RA isthmus line and demonstration of bidirectional block.

FOLLOW UP Patients will be followed up at 3, 6, and 12 months.

DETAILED DESCRIPTION:
FOLLOW UP

Patients will be followed up at 3, 6, and 12months with:

* clinical visit, symptoms questionnaire, electrocardiogram (ECG), ECG Holter (3, 6, and 12 months);
* trans-thoracic echocardiogram (only at 12months);
* Three-dimensional late gadolinium enhancement cardiac magnetic resonamce - 3D LGE- CMR (if possible, only at 6 months); exercise cardiopulmonary test (only pre-ablation and at 6 months).

SAFETY REPORTING RECORDING ADVERSE EVENTS (AES) All Adverse Events will be recorded in the hospital notes and Case Report Form (CRF).

If the Investigator suspects that the disease has progressed faster due to the administration of the study treatment/procedure, then he/she will report this as an unexpected adverse event to the Sponsor and the REC.

THE TYPE AND DURATION OF THE FOLLOW-UP OF SUBJECTS AFTER AES The type and duration of follow-up care for subjects following an AES will be as follows: 6-12 months following pulmonary vein stenosis, phrenic nerve palsy, valve damage, and atrio-oesophageal fistula (if operated); 3-6 months following vascular complications or pericardial effusion (usually these complications are promptly treated without major long term consequence).

PREGNANCY Pregnant patients will be excluded from the study. However, if pregnancy occurs after inclusion into the study, investigators will record and notify pregnancies occurring during the study period to the Sponsor.

Follow-up of pregnant subject:

* No further ablation procedure will be undertaken during the pregnancy period in order to avoid radiation exposure and hazards to the foetus.
* Medication contraindicated during pregnancy will be withdrawn.
* Anticoagulation treatment with Warfarin will be discontinued during the first and the third trimester and replaced with subcutaneous injections of low molecular weight heparin.
* No additional investigations involving radiation exposure such as computed tomography (CT), X ray will be performed, unless clinically urgent.

Follow-up of child born to a pregnant trial subject, including male trial subject who is the partner of the pregnant woman:

Children born to a pregnant subject are unlikely to be affected by the participation of the parent in the study. For safety reasons, a specialised paediatric team will follow children for 1 year.

ANNUAL PROGRESS REPORTS (APRS) The Chief Investigator (CI) will prepare the APR for the study. It will be reviewed by the Research Office (RO) and sent to the regulatory ethic committee (REC) by the CI within 30 days of the anniversary date on which the favorable opinion was given by the REC, and annually until the study is declared ended.

REPORTING URGENT SAFETY MEASURES The Sponsor and/or the Investigator may take appropriate urgent safety measures in order to protect the subjects of a clinical study against any immediate hazard to their health or safety. If safety measures are taken, REC approval is not required before the measure is taken.

The Investigator will immediately and in any event no later than 3 days from the date the measures are taken, give written notice to the REC and the study Sponsor of the measures taken and the circumstances giving rise to those measures.

In order to prevent any delays in the reporting timelines the Sponsor has delegated this responsibility to the CI/Principal Investigator (PI). Therefore, the CI/PI must report any urgent safety measures to the REC directly, and in parallel to the Sponsor. The REC coordinator will acknowledge receipt of urgent safety measures within 30 days.

DATA MANAGEMENT AND QUALITY ASSURANCE CONFIDENTIALITY All data will be handled in accordance with the Data Protection Act 1998, NHS Caldecott Principles, The Research Governance Framework for Health and Social Care, 2nd Edition (2005), and the condition of the REC approval.

The Case Report Forms (CRFs) will not bear the subject's name or other personal identifiable data. The subject's initials, Date of Birth (DOB) and study Identification Number (ID), will be used for identification.

DATA COLLECTION TOOL Case Report Forms (CRF) will be designed by the CI and the final version will be reviewed and discussed with the study Sponsor. All data will be entered legibly in black ink with a ball-point pen. If the Investigator makes an error, it will be crossed through with a single line in such a way to ensure that the original entry can still be read. The correct entry will then be clearly inserted. The amendment will be initialled and dated by the person making the correction immediately. Overwriting or use of correction fluid will not be permitted.

It is the Investigator's responsibility to ensure the accuracy of all data entered and recorded in the CRFs. The Delegation of Responsibilities Log will identify all trial personnel responsible for data collection, entry, handling and managing the database.

Data will be firstly recorded into source documents (i.e medical notes) (medical history, baseline investigations) and then recorded onto the CRF (with the addition of the procedure specific data).

Methods used to maximise completeness of data will include telephoning subjects who have not attended the planned follow-up visit.

DATA HANDLING AND ANALYSIS

* Excel software will be used for data entry.
* In order to ensure validity and quality of data the study investigators will use cross validation
* Data will be stored and backed up on 2 additional hard drives on two different sites in order to allow recovery of data in case of a disaster such as fire/flooding/ theft. The PI and their collaborators/co-workers will be responsible for data entry and quality of data collection. Analysis will be performed by the study investigators and reviewed independently of data entry by the statistical team.
* Every patient will receive a numerical patient identifier and all data that is transferred outside the primary hospital will exclusively be identified by this study number.
* The study database will be held at the Biomedical Research Unit (BRU) server at the Royal Brompton Hospital.

ARCHIVING ARRANGEMENTS The study documents (including the Study Master File (SMF), Case Report Forms (CRFs), Informed Consent Forms along with the study database) will be kept for a minimum of five years. They will be stored in locked offices within the Royal Brompton and Harefield NHS Foundation Trust (RB&HFT). The CI is responsible for the secure archiving of study documents. The study database will also be kept electronically on the RB&HFT computer network, for a minimum of five years.

The approved repository for longer retention of local materials for studies that involve RB&HFT patients is Box-It Storage UK. The study documentation will be prepared for archiving by the research team in line with the Research Office Archiving Standard Operating Procedures (SOP) and the transfer will be arranged by the Research Office.

Patient anonymised data may be exported for the purpose of offline review and to perform the image merge as part of the study and also to further develop the technology.

STATISTICAL ANALYSIS This is a feasibility pilot study, which will test the feasibility of AF mapping with Acutus system and catheter ablation in patients with HCM and paroxysmal or persistent AF (time in persistent AF < 12 months duration). Therefore, no power calculation has been done and the number of patient recruited will be of 20 which are deemed sufficient by the Chief Investigator and Co-PIs on a clinical basis.

The estimated recruitment period for the trial will be of 6 months. We estimate that this sample size is attainable in practice, as the number of AF ablation procedures per year performed within each Trust is around 400. The study investigators also included patients with previous AF ablation in order to maximise chances of recruitment. This pilot is performed with the intention to plan a prospective multi-operator/multicentre trial which is adequately powered.

The study investigators will aim to compare the procedure parameters as well as the outcome of this trial to age & gender matched procedures of the same operator from the last 5 years' database.

STATISTICAL ANALYSIS PLAN Descriptive statistic data with regard to baseline and procedural variables will be reported; continuous variables will be expressed by mean ± standard deviation or median and interquartile range (25th, 75th percentile), depending on the normality of distribution; categorical variables will be summarized by frequencies and percentages. The outcome of radiofrequency ablation on the entire cohort of patients will be presented in the form of percentage of patients free from symptomatic or documented arrhythmia or with only mild symptoms related to arrhythmia recurrence. Results will be reported separately for 3, 6 and 12month visit.

Depending on the severity of symptoms and documentation of tachycardia during follow-up, patients will be divided into two groups (success/recurrence). Baseline characteristics and procedural variables will be compared between these two groups by student t-tests, Mann Whitney U tests, or Fisher's exact test where appropriate in order to identify those variables associated with better mid/long term outcomes. A two-tailed p value <0.05 will be considered statistically significant. Intra-patient improvement from baseline to 12 months follow-up visit will be assessed by McNemar's test. Freedom from AF will be assessed as a time dependant variable using Cox proportional hazard models.

To judge if ablation strategy using Acutus mapping system is as successful in achieving the clinical endpoint, the study investigators will compare the procedure parameters as well as the outcome of this trial to age & gender matched procedures of the same operator from the last 5 years' database.

To measure the strength of association between the acute successes (SR at the end of the ablation), 3, 6 and 12-month outcomes, a McNemar test will be performed. Data will be analysed using SPSS version 18 (IBM Corporation).

RANDOMISATION The subjects will be randomly assigned to one of the two procedures using a computer programme that provides a sequence of the procedures randomly permuted in blocks of constant or varying size. For this study a constant block size will be used.

COMMITTEES INVOLVED IN THE STUDY Trial Management Group (TMG) - normally includes those individuals responsible for the day-to-day management of the trial, such as the CI, statistician, trial manager, research nurse, data manager. The role of the group is to monitor all aspects of the conduct and progress of the trial, ensure that the protocol is adhered to and take appropriate action to safeguard participants and the quality of the trial itself.

MONITORING AND AUDITING The requirement for study monitoring or audit will be based on the internal Research Office (RO) risk assessment procedure and applicable Standard Operating Procedures (SOPs). It is the responsibility of the RO to determine the monitoring risk assessment and explain the rationale to the study research team. Monitoring support will be provided by the Sponsor, Spectrum Dynamics, as required.

Study monitoring and/or audit will be discussed with the CI before arrangements are made to conduct the visit.

DIRECT ACCESS TO SOURCE DATA The Investigator(s)/institution(s) will permit trial-related monitoring, audits, REC review, and regulatory inspection(s), providing direct access to source data/documents. Trial participants are informed of this during the informed consent discussion. Participants will consent to provide access to their medical notes.

FINANCE The therapeutic procedure follows the normal clinical pathway for treatment of atrial fibrillation. The additional cost incurred due to the participation in the HCM-AF ablation with Acutus protocol per patient will be sponsored by Acutus Medical.

INSURANCE AND INDEMNITY NHS bodies are liable for clinical negligence and other negligent harm to individuals covered by their duty of care. NHS Institutions employing researchers are liable for negligent harm caused by the design of studies they initiate. The provision of such indemnity for negligent harm should be stated to the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal or persistent AF (time in persistent AF < 12 months duration) including re-ablations
2. Able to give written informed consent
3. Age >18 years old and ≤ 80 years
4. Fulfil established clinical criteria for diagnosis of HCM and catheter ablation of atrial fibrillation
5. Normal LV ejection fraction and no evidence of other significant structural heart disease

Exclusion Criteria:

1. Reversible causes of AF/flutter/tachycardia
2. Recent cardiovascular event including TIA
3. Intolerance or unwillingness to oral anticoagulation with Warfarin or NOAC
4. Bleeding disorder
5. Contraindication to CT or CMR scan
6. Presence of intra-cardiac thrombus
7. Vascular disorder preventing access to femoral veins
8. Cardiac congenital abnormality different from HCM
9. Severe, life threatening non cardiac disease
10. Active malignant disease and recent (<5 years) malignant disease
11. Presence of ASD or PFO closure device
12. Previous ASD or PFO surgical closure
13. Unable or unwilling to comply with F/U requirements
14. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy to achieve SR defined as time (in minutes) to termination of AF into stable SR | 12 months
  • Assessment on efficacy of ACUTUS mapping system guided AF ablation in HCM patients using a double-arm study design. Time to termination of AF to SR
Acute procedural safety assessed by incidence (number and type) of acute procedure-related Adverse Events | 12 months
  • Absence of acute adverse events due to the use of ACUTUS mapping system during AF ablation
Chronic procedural safety assessed by incidence (number and type) of chronic procedure-related Adverse Events | 12 months
  • Evidence of chronic adverse events due to the use of ACUTUS mapping system guided catheter ablation during the 12 months F/U period
Overall safety of the entire mapping and ablation strategy defined by incidence (number and type) of acute and chronic Adverse Events, differentiated into those related to the mapping system (ACUTUS) and those related to the ablation procedure | 12 months
  • Safety endpoint of the entire mapping and ablation strategy

SECONDARY OUTCOMES:
Overall RF time delivered till SR | 12 months
  • RF time to termination of AF to AT
clinical long term outcome | 12 months
  • Freedom from AF/flutter/tachycardia (> 30 sec) at the end of the 12 months F/U period
Time to first recurrence | 12 months
  • Time to first recurrence of AF/flutter/tachycardia (> 30 sec)
Clinical outcome including drugs | 12 months
  • Freedom of AF/flutter/tachycardia on previously failed anti-arrhythmic medication

IPD SHARING:
Plan to Share IPD: No